CLINICAL TRIAL: NCT00730509
Title: Preliminary Evidences of Active Form of Folic Acid and Vitamin B12 Supplementation to Ameliorate Cell Membrane in Children With Cystic Fibrosis
Brief Title: Effects of 5-Methyltetrahydrofolate and Vitamin B12 Supplemetation on Red Cell Membrane in Children With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Prof. Lisa Maria Bambara, Verona University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UNIVR_REUM_01
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-05

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; folate; vitamin B12
MeSH Terms: conditions — Cystic Fibrosis | interventions — 5-methyltetrahydrofolate; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: 5-methyltetrahydrofolate and vitamin B12 — children with cystic fibrosis were supplementated for 6 months with 5-MTHF, 7,5 mg/day ; vitamin B12, 0,5 mg/day

SUMMARY:
The purpose of this study is to determine whether 5 - methyltetrahydrofolate and vitamin B12 supplementation can ameliorate cell plasma membrane features in pediatric patients with cystic fibrosis

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is one of the most common fatal autosomal recessive disorders in the Caucasian population caused by mutations of gene for the cystic fibrosis transmembrane conductance regulator (CFTR). New experimental therapeutic strategies for CF propose a diet supplementation to affect the plasma membrane fluidity and to modulate the cellular amplified inflammatory response in CF target organs. Red blood cells (RBCs) were used to investigate plasma membrane, because RBCs share lipid, protein composition and organization with other cell types.

ELIGIBILITY:
Inclusion Criteria:

* cystic fibrosis

Exclusion Criteria:

* diabetes
* chronic infections of the airways
* regular antibiotics intake

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2004-04; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
We evaluated membrane protein oxidative damage of red cells | 6 months

SECONDARY OUTCOMES:
we evaluated cation transport pathways of red cells | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M. Bambara, MD, Study Director — Verona University
Locations (1):
- Verona University, Verona, Italy

REFERENCES:
- [Background] Scambi C, Guarini P, De Franceschi L, Bambara LM. Can 5-methyltetrahydrofolate modify the phospholipid fatty acid pattern in cystic fibrosis pediatric patients? J Cyst Fibros. 2006 Aug;5(3):197-9. doi: 10.1016/j.jcf.2006.01.006. Epub 2006 Mar 3. PMID 16516563
- [Derived] Scambi C, De Franceschi L, Guarini P, Poli F, Siciliano A, Pattini P, Biondani A, La Verde V, Bortolami O, Turrini F, Carta F, D'Orazio C, Assael BM, Faccini G, Bambara LM. Preliminary evidence for cell membrane amelioration in children with cystic fibrosis by 5-MTHF and vitamin B12 supplementation: a single arm trial. PLoS One. 2009;4(3):e4782. doi: 10.1371/journal.pone.0004782. Epub 2009 Mar 11. PMID 19277125